CLINICAL TRIAL: NCT04597515
Title: Reduction of Breast Enlargement Using the Da Vinci Xi Robot
Acronym: R-HTM-R
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Hôpital Privé d'Antony - Dr Dunet (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2019-A01199-48
Record Dates: First submitted 2020-06-02; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Breast Hypertrophy
Keywords: breast reduction; perimammary
MeSH Terms: conditions — Gigantomastia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot Reduction (Experimental): The project consists in removing a breast disc at the base, causing a circular sagging skin cut of 2 to 3 cm .
  Interventions: Procedure: Robot Breast reduction surgery

INTERVENTIONS:
Procedure: Robot Breast reduction surgery — Breast reduction surgery, using a robot by removing a breast disc at the base

SUMMARY:
Breast enlargement reductions are frequent interventions. One of the main issue associated with this surgery remains the ransom scar, wide at the periareolar level, vertical at the subareolar level and in the submammary groove.

The expected result is to achieve a reduction in breast enlargement with no visible scar using Da Da Vinci Xi robot.

DETAILED DESCRIPTION:
Breast enlargement reductions are frequent interventions. One of the main issue associated with this surgery remains the ransom scar, wide at the periareolar level, vertical at the subareolar level and in the submammary groove. In addition, this intervention remains subject to the vagaries of hypertrophic or even keloid scarring, especially in young women.

The current research project is based on the hypothesis that the same technique could be used in the context of a reduction of breast enlargement on a smaller surface allowing the determination of a perimammary "halo" of scar retraction. The project consists in removing a breast disc at the base, thus causing a sagging skin cut of 2 to 3 cm but this time, circular.

The expected result is to achieve a reduction in breast enlargement with no visible scar, using Da Vinci Xi robot.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18
* Category 1 or 2 according to the classification of Regnault
* Breast size cup c or more
* Areola "looking in front", ie a distance between point A (at noon at the top of the areola) at the mid-sternal point of about 16 cm to 24 cm
* Ptosis (distance between the lowest part of the breast and the furrow under the breast) to a maximum of 7cm (measurement in sitting position)
* Expected correction of ptosis by half with reduction of 1 to 3 cup sizes
* Good quality thick skin
* Affiliated patient or beneficiary of a social security scheme
* Patient requesting breast reduction
* Patient who signed free and informed consent

Exclusion Criteria:

* Areola "look down"; point A more than 25 cm
* Ptose greater than and equal to 8 cm
* Thin skin
* Smoker
* Patient on anti-coagulant
* Patient participating in another clinical study
* Protected patient: adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision;
* Pregnant, lactating woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Visible Scare | 3 months
  The main judgment criterion for the scar balance will be a photograph of the breasts at 3 months to describe the number of visible scars. Aspect and position.

SECONDARY OUTCOMES:
Efficacity of the reduction (weight) | day of surgery
  - The weight of the exeresis (more than 300g per side which corresponds according to calculation to a gland disc about 2 cm thick on an extended conical breast of 13cm for the base)
Intensity of Back Pain | 3 months
  The pain score on the EVA scale (score from 0 no pain to 10 max pain) will be described
Skin retraction | at 3 months
  - Post-operative skin retraction

OTHER OUTCOMES:
Visible scare number | 1 year
  number of visible scare based on photos analysis

CONTACTS AND LOCATIONS:
Overall Officials: Eric Dunet, Dr, Principal Investigator — Ramsay santé
Locations (1):
- Hôpital Privé d'Antony, Antony, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided